CLINICAL TRIAL: NCT01669525
Title: Placental Growth and Maternal Serum Biomarkers in the Prediction of Adverse Pregnancy Outcome
Brief Title: Placental Growth and Adverse Pregnancy Outcomes
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 811129
Record Dates: First submitted 2012-08-15; First posted 2012-08-21 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Hypertension Induced by Pregnancy; Pre-Eclampsia; IUGR
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal serum will be collected. Placental biopsies may be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Singleton pregnancies presenting to the Genetic Counselor for Sequential Screening prior to 14 weeks gestation.

SUMMARY:
The purpose of this study to determine if measurement of maternal serum biomarkers and evaluation of the placenta by ultrasound can improve prediction of adverse pregnancy outcomes.

DETAILED DESCRIPTION:
The placenta is known to play a vital role in maintaining a healthy pregnancy. Placental dysfunction is believed to be a driving factor in a variety of adverse obstetric outcomes, including fetal growth restriction and preeclampsia. Advances in 3D ultrasound have allowed for measurement of placental volumes during pregnancy. It may be that quantitative assessment of early placental growth can help identify pregnancies at risk for adverse outcome. Furthermore, various novel serum analytes have been proposed as predictors of adverse outcome. The investigators seek to prospectively measure placental volume and diameter at 11-14 weeks and 18-24 weeks to determine if placental growth can predict adverse outcome. In addition, the investigators seek to investigate the relationship between placental growth and serum levels of various biomarkers to see if improved detection of adverse outcome can be achieved.

ELIGIBILITY:
Inclusion Criteria:

* All singleton gestations presenting for Sequential Screen testing at HUP
* patients competent to provide verbal informed consent

Exclusion Criteria:

* Multiple gestations
* patients not competent to provide informed consent
* patients found to be too late for the Sequential Screen
* pregnancy losses 20 weeks gestation
* major fetal anomalies
* patient delivering outside of the UPHS

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Singleton pregnancies presenting for Sequential Screen prior to 14 weeks gestation
Sampling Method: Non-Probability Sample
Enrollment: 1043 (Actual)
Dates: Start 2009-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Small for gestational birth weight (SGA-dichotomous) | from 11-14 weeks in pregnancy until delivery (approximately 40 weeks)
  Neonatal weight and length are recorded at birth. This information will be retrieved from the medical record post partum.

SECONDARY OUTCOMES:
Includes a composite adverse outcome defined by any of the following: SGA, pre-eclampsia, or perinatal death. | post partum
  Information about pregnancy outcomes will be retrieved from the maternal and neonatal medical record post partum.

CONTACTS AND LOCATIONS:
Overall Officials: Nadav Schwartz, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States